CLINICAL TRIAL: NCT01603212
Title: Systemic Therapy of Metastatic Melanoma With Multidrug Regimen Including Interferon, Interleukin-2 and BRAF Inhibitor
Brief Title: Systemic Therapy With Interferon, Interleukin-2 and BRAF Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0847; NCI-2012-02759 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic melanoma; Advanced melanoma; Vemurafenib; PLX4032; RO5185426; IL-2; Interleukin-2; Aldesleukin; Proleukin; Interferon Alfa-2b; Intron A
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Interleukin-2; aldesleukin; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vemurafenib + IL-2 + Interferon Alfa-2b (Experimental): Starting dose of Vemurafenib 720 mg by mouth twice daily. Three dose levels of Vemurafenib evaluated in combination with interferon and IL-2. These doses are 480 mg, 720 mg and 960 mg. IL-2 given by continuous venous infusion at starting IL-2 dose of 7 million IU/m2 daily for 4 days (total of 96 hours, days 2-5) starting day 2. IL-2 dose levels are 5MU/m2/day, 7MU/m2/day and 9MU/m2 day. Doses of interferon remain constant at 5 MU/m2 subcutaneously daily for 5 days starting Day 1.
  Interventions: Drug: Vemurafenib; Drug: IL-2; Drug: Interferon Alpha-2b

INTERVENTIONS:
Drug: Vemurafenib — Phase I Starting dose: 720 mg by mouth twice a day for a 21 day cycle.
  Phase II Starting dose: Maximum tolerated dose (MTD) from Phase I.
  Other Names: PLX4032; RO5185426
Drug: IL-2 — Phase I Starting Dose: 7 million IU/m2 by vein on Days 2 - 5 of a 21 day cycle.
  Phase II Starting Dose: Maximum tolerated dose (MTD) from Phase I.
  Other Names: Interleukin-2; Aldesleukin; Proleukin
Drug: Interferon Alpha-2b — 5 million U/m2 subcutaneously on Days 1 - 5 of a 21 day cycle.
  Other Names: Intron A

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of vemurafenib and Aldesleukin (interleukin-2) that can be given in combination with interferon alfa-2b in patients with advanced or metastatic melanoma. The safety of this combination will also be studied.

The goal of Phase II is to learn if this study drug combination can help to control advanced or metastatic melanoma.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of 6 participants will be enrolled in the Phase I portion of the study and up to 53 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of vemurafenib and aldesleukin you receive will depend on when you joined this study. The first group of participants will receive the lowest dose levels of vemurafenib and aldesleukin. Each new group will receive a higher dose of vemurafenib or aldesleukin than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable doses of vemurafenib and aldesleukin are found.

If you are enrolled in the Phase II portion, you will receive vemurafenib and aldesleukin at the highest doses that were tolerated in the Phase I portion.

All participants will receive the same dose level interferon alfa-2b.

Study Drug Administration:

Each study cycle is 21 days.

You will take vemurafenib by mouth twice a day (1 time in the morning and 1 time in the evening) every day of each study cycle. Vemurafenib can be taken with or without food. If you miss a scheduled dose of vemurafenib, do not try to "make up" the dose by taking 2 doses at the next scheduled dosing time. Continue taking the study drug as scheduled.

You will receive aldesleukin by vein over 96 hours on Days 1-4 of each study cycle.

To receive aldesleukin, you will have a central venous catheter (CVC) inserted, if you do not already have one. A CVC is a sterile flexible tube that will be place into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

You will receive interferon alfa-2b as an injection under your skin on Days 1-5 of each study cycle.

Supportive Drugs:

You will be given other drugs to help lower the risk of side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

The following tests and procedures will be performed:

On Day 1 (+/- 3 days) of each cycle:

* Your performance status will be recorded.
* Your vital signs will be measured.
* You will be asked about any drugs you may be taking and any side effects you may have had.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.
* You will have an EKG.

Your skin will be checked for non-melanoma skin cancers on Day 1 of Cycle 1 (+/- 3 days) and then every 3 cycles.

Blood (about 1 teaspoon) will be drawn for routine tests on Days 1, 8, and 15 of each cycle. On Day 1 of each cycle, some of this blood will be used to check your liver and kidney function.

At the end of each cycle (Day 21), you will have a physical exam, including measurement of your weight. Any tumor that can be felt with the hands will be measured with measuring tape during the physical exam to see if it has changed size.

On Day 21 (+/- 7 days) of every 2 cycles, you will have a chest x-ray and a CT or MRI scan to check the status of the disease.

Anytime the doctor thinks it is needed, photos of any skin lesions you have will be taken. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are lesions on your face.

Length of Study:

You may take the study drug combination for as long as the doctor thinks you are benefitting. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit

Within 14 days after you stop taking the study drug combination, the following tests and procedures will be performed:

* Your performance status will be recorded.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any drugs you may be taking and any side effects you may have had.

vBlood (about 2 tablespoons) will be drawn for routine tests.

° If the doctor thinks it is needed, you will have a CT or MRI scan.

Follow-Up Every 3 months for up to 3 years, you will be contacted by phone or during a clinic visit to see how you are doing. The phone call should last about 5 minutes.

This is an investigational study. Vemurafenib, interferon alfa-2b, and Aldesleukin are FDA approved and commercially available to treat metastatic cancer. Giving these drugs in combination is investigational. The study doctor will tell you how the study drugs are designed to work.

Up to 71 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III skin or mucosal melanoma are eligible if they have BRAF mutation affecting the V600 site, as determined by a chemiluminescence immunoassay analyzer (CLIA)-certified assay. Mutation testing of archival tumor tissue is acceptable, or it may be performed on new biopsy. If a new biopsy is performed for testing, biopsy of a metastasis is preferred to biopsy of a primary tumor.
2. Patients must have at least one bidimensionally measurable lesion. If this is a cutaneous lesion it must be at least 10 mm by caliper measure. If it is a visceral or nodal or soft tissue lesion, it must be clearly measurable > 20 mm with conventional techniques or > 10 mm with spiral CT scan. Bone lesions are not considered measurable.
3. Phase I: Patients with prior therapy who do not have alternative treatment of higher priority will be eligible. Phase II: the patient may have been treated with cytotoxic drugs or targeted therapies for metastatic disease but not with IL-2, interferon and BRAF inhibitor drugs. Adjuvant interferon will be permitted. Prior radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity. Prior chemotherapy is permitted provided the patient has a 21 day wash out period and the patient has fully recovered from its toxicity.
4. Patients between 18 years of age and 65 years of age with an Eastern Cooperative Oncology (ECOG) performance status of 0, 1 or 2 will be eligible.
5. They should have normal blood counts with a white blood cell count (WBC) count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3 and have no impairment of renal function (serum creatinine less than 1.1 mg/dl for females and less than 1.4 mg/dl for males), hepatic function (serum bilirubin level of less than 1.2 mg/dl) and no evidence of significant cardiac or pulmonary dysfunction.
6. They should have no significant intercurrent illness such as an active infection associated with fever lasting more than 24 hours requiring antibiotics, uncontrolled psychiatric illness, hypercalcemia (calcium greater than 11 mg), active GI bleeding, myocardial disease with corrected QT interval (QTC) interval > 480 on baseline ECG or history of rheumatoid arthritis.
7. Females of child-bearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods( abstinence, intrauterine device, oral contraceptive or double barrier devices) and must have a negative serum or urine pregnancy test within 72 hours prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.

Exclusion Criteria:

1. Patients with uveal melanoma.
2. Patients with bone metastases only.
3. Patients with brain metastases unless all of their metastatic brain lesions have been resected or treated with stereotactic radiotherapy with gamma rays and they are off corticosteroids. Patient should not have significant brain edema. Patients with spinal cord compression and leptomeningeal disease. No major surgery or radiation therapy within 21 days before starting treatment.
4. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (Ejection Fraction less than 50%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients will be evaluated by the investigator or his designee.
5. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of forced expiratory volume at one second (FEV1) to less than 65 % of predicted normal values.
6. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
7. Patients who are unable to return for follow-up visits as required by this study.
8. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 3 years and uncertainty about the histological nature of the metastatic lesions. Cases with other types of malignancies should be reviewed and decided by the PI of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Vemurafenib in Combination With Interferon Alpha 2b and IL-2 | 21 days
  Maximum tolerated dose (MTD) defined as highest dose studied in which incidence of dose limiting toxicity (DLT) was less than 33%. DLT defined as any grade 3 or 4 non-hematological toxicity excluding manageable N/V, diarrhea and fatigue and manageable/replaceable grade 3 or 4 electrolyte abnormalities, and appearance of new squamous cell skin cancers. Toxicity that may result in delaying next course for more than 3 weeks. Any grade 4 neutropenia more than 7 days duration or Grade 4 thrombocytopenia lasting more than 7 days.
Progression-Free Survival (PFS) | 6 months
  Progression-free survival estimated using the method of Kaplan-Meier. It will be determined from the start of the study until disease progression or death, whichever is first.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N. Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org